CLINICAL TRIAL: NCT06907199
Title: A Multicentric Randomized Trial of Daily Nitrofurantoin Versus Bladder Fulguration Plus Daily Nitrofurantoin for the Long-term Management of Cystitis in Women With Recurrent Urinary Tract Infections
Brief Title: Daily Nitrofurantoin Versus Bladder Fulguration Plus Daily Nitrofurantoin for Women With Recurrent Urinary Tract Infections
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: University of Texas (Other); National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Philippe Zimmern, Professor of Urology, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU-2024-1187; 1R01DK140224-01A1 (NIH)
Record Dates: First submitted 2025-03-24; First posted 2025-04-02 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Recurrent UTIs; Cystitis Recurrent
Keywords: bladder fulguration; Nitrofurantoin; long-term managenent of cystitis; Recurrent UTI; chronic UTI
MeSH Terms: conditions — Urinary Tract Infections | interventions — Diathermy; Nitrofurantoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Nitrofurantoin (NF) daily antibiotic prophylaxis (Active Comparator): Nitrofurantoin (NF) daily antibiotic prophylaxis given daily for 6 months.
  Interventions: Drug: Nitrofurantoin (NF)
- Nitrofurantoin (NF) daily antibiotic prophylaxis plus electrofulguration (EF) (Experimental)
  Interventions: Procedure: Electrofulguration (EF); Drug: Nitrofurantoin (NF)

INTERVENTIONS:
Procedure: Electrofulguration (EF) — Nitrofurantoin (NF) daily antibiotic prophylaxis for 6 months plus Electrofulguration.
  Other Names: fulguration
  Arms: Nitrofurantoin (NF) daily antibiotic prophylaxis plus electrofulguration (EF)
Drug: Nitrofurantoin (NF) — Nitrofurantoin (NF) daily antibiotic prophylaxis given daily for 6 months.

SUMMARY:
The goal of this clinical trial is to learn if the drug Nitrofurantoin (NF) taken as a daily antibiotic, works to treat cystitis compared to electrofulguration (EF) and Nitrofurantoin (NF) daily antibiotic.

DETAILED DESCRIPTION:
This is a study for women age 18 -85 with a well-documented history of rUTI (recurrent urinary tract infection) for at least one year. This randomized multicentric clinical trial will determine the efficacy of conventional 6 months Nitrofurantoin (NF) daily antibiotic prophylaxis alone versus electrofulguration (EF) associated with a 6 months NF daily antibiotic prophylactic course for early stages of chronic cystitis (stages 1 and 2) as determined on office cystoscopy.

This study will ask the participant (n=104) to return to the Urology clinic at UT Southwestern Medical Center (n=52) or The University of Kansas Medical Center (n=52) for a total of 8 compensated visits throughout 30 months after the start of this randomized trial to make sure that the treatment worked well for them.

ELIGIBILITY:
Inclusion Criteria:

* Females 18 to 85 years old with at least a 1-year history of culture documented uncomplicated rUTI.
* Diagnosis of rUTI, defined as ≥ 3 symptomatic UTIs in 12 months or ≥ 2 in 6 months.
* Currently free from a UTI determined based on absence of symptoms as determined by the UTI symptom assessment questionnaire and negative urine culture (<10^3 colony forming units per ml of urine).
* A negative upper and lower urinary tract evaluation, including pelvic examination for pelvic organ prolapse (less than or equal to stage 2), measurement of post-void residual (less than 50 ml), and imaging (which may include renal ultrasound and standing voiding cystourethrogram) to exclude kidney stone, hydronephrosis, reflux, or urethral diverticulum.
* Office cystoscopy documenting stages 1 or 2 of chronic cystitis.
* Likely to stay in the geographic region for the duration of the study.
* ASA class II or less.

Exclusion Criteria:

* Patients on antibiotics at baseline (i.e., suppressive therapy or antibiotic therapy for non-urinary infections).
* Patients on self-start therapy (i.e., taking antibiotics upon start of urinary symptoms concerning for UTI).
* Patients on prophylactic antibiotics started in the last 3 months and unwilling to discontinue, or intention to start in the next 12 months.
* Complicated UTIs, including neurogenic bladder condition (i.e., multiple sclerosis, Parkinson's disease, spinal cord injury), bladder augmentation, or urinary diversion.
* Patients with urinary catheters (including indwelling Foley, intermittent catheterization, and suprapubic catheters).
* Uncontrolled diabetes (HbA1c >9).
* Pregnancy
* Allergy or resistance to Nitrofurantoin.
* Chronic lung or liver condition precluding the use of Nitrofurantoin, including abnormal chest X ray or elevated liver function tests.
* Chronic renal insufficiency (creatinine over 1.5 g/dl or GFR less than 40) precluding the use of Nitrofurantoin.
* History of chronic diarrhea requiring regular therapy.
* Patients with psychosis, dementia, swallowing disorders, or any other ability to take Nitrofurantoin reliably at home.
* BMI over 40.
* Use of Uromune or other vaccine approaches to reduce rUTI episodes
* Participation in a research study involving an investigational product in the past 12 weeks.
* Patients receiving phage therapy.
* Current diagnosis of interstitial cystitis.
* Patients with medical conditions requiring excessively large amounts of fluid intake.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Biologically born female
Enrollment: 104 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2028-07-01 (Estimated); Study Completion 2029-01-30 (Estimated)

PRIMARY OUTCOMES:
Treatment of cystitis with NF vs EF+NF | Baseline to 30 months after enrollment to completion of study
  Rate of culture documented symptomatic UTIs following the completion of each 6-month study arm intervention. Specifically, from 6 to 18 months (first year) after the completion of the original intervention and, 18 to 30 months (second year).

SECONDARY OUTCOMES:
No recurring cystitis | Baseline to 30 months after enrollment to completion of study
  Comparison of patient characteristics between the two enrolling institutions.
Rate comparison of culture-documented breakthrough | Baseline to 30 months after enrollment to completion of study
  Rate of culture-documented breakthrough UTIs between the two treatment arms.
Rate of multi-drug resistant organisms | Baseline to 30 months after enrollment to completion of study
  Rate of urine cultures showing multi-drug resistant organisms in each treatment arm.
Rate of non-urine culture | Baseline to 30 months after enrollment to completion of study
  Rate of non-urine culture documented symptomatic UTI episodes for 12 months and 24 months following end of treatment arms, as determined by the Urinary Tract Infection Symptom Assessment (UTISA) (a total score of 3 or higher, or any individual score of 2 or 3) between the two treatment arms.
Rate of behavior changes | Baseline to 30 months after enrollment to completion of study
  Rate of behavior changes in both groups (fluid increases or use of non-antibiotic therapies, e.g., cranberry, D-mannose, urinary analgesics, hormonal therapy) in each treatment arm.
Rate of score differences in symptoms and quality of life | Baseline to 30 months after enrollment to completion of study
  Rate of score differences in patient symptoms and quality of life assessments using validated questionnaires- the Urinary Tract Infection Symptom Assessment (UTISA), Urinary Distress Inventory, Short Form (UDI-6), and Quality of Life scale (QoL) by Visual Analogue Scale (VAS) between both treatment arms.
Rate of UTI episodes | Baseline to 30 months after enrollment to completion of study
  Rate of UTI episodes (after first and second year of the completion of the intervention) compared to the rate of UTI episodes prior to the start of study

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - The University of Kansas, Kansas City, Kansas
  - UT Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Undecided